CLINICAL TRIAL: NCT04735965
Title: Comparison of Dexmedetomidine and Meperidine for the Prevention of Shivering Following Coronary Artery Bypass Graft: Study Protocol of a Randomized Controlled Trial
Brief Title: Comparison of Dexmedetomidine and Meperidine for the Prevention of Shivering Following Coronary Artery Bypass Graft
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMCABG
Record Dates: First submitted 2021-01-24; First posted 2021-02-03 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Coronary Artery Disease; Postoperative Shivering
Keywords: Shivering
MeSH Terms: conditions — Coronary Artery Disease | interventions — Dexmedetomidine; Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine
- Meperidine group (Active Comparator)
  Interventions: Drug: Meperidine
- Control group (Placebo Comparator)
  Interventions: Drug: Placeb

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine would be intravenously infused at a dose of 1μg/kg over 15 minutes 30 min before the end of surgery
  Arms: Dexmedetomidine group
Drug: Meperidine — Meperidine would be intravenously injected at a dose of 0.5mg/kg 30 min before the end of surgery
  Arms: Meperidine group
Drug: Placeb — Equal volume of normal saline to dexmedetomidine and meperidine group.
  Arms: Control group

SUMMARY:
This study aims to compare the effects of dexmedetomidine and meperidine on the incidence of shivering in patients undergoing CABG.

DETAILED DESCRIPTION:
Shivering is a common complication in the postoperative period. The incidence of shivering has been reported to range from 5% to 65% under general anesthesia and as 33% during epidural anesthesia. Shivering can increase perioperative risk in patients. Both dexmedetomidine and meperidine are effective agents for the prevention of postanesthetic shivering. However, few studies have compared the anti-shivering effects of different agents following coronary artery bypass graft (CABG). This study aims to compare the effects of dexmedetomidine and meperidine on the incidence of shivering in patients undergoing CABG.

ELIGIBILITY:
Inclusion Criteria:

(1) aged between 18 and 75 years, (2) undergoing elective CABG, (3) ASA grade of II-IV, and (4) in accordance with ethical guidelines, patients must voluntarily participate in the trial and sign the informed consent for the clinical study.

Exclusion Criteria:

(1) patients with neurological or psychiatric disorders, (2) hepatic and renal dysfunction, (3) severe hyperthyroidism or hypothyroidism, (4) a body temperature greater than 38 °C or less than 36 °C, (5) postoperative hemodynamic instability, (6) preoperative use of a left ventricular assistance device, (7) pa severe diabetic complications (diabetic ketoacidosis, hyperosmolar coma, various infections, diabetic nephropathy), (8) participation in other clinical studies within the past 3 months, (9) acute or chronic pain, (10) addiction to opioids, (11) drug abuse, (12) pain management, and (13) neuromuscular disease, (14) on-pump CABG.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative shivering | Within postoperative 24 hours
  The incidence and severity of postoperative shivering and the rescue treatment

SECONDARY OUTCOMES:
Times of postoperative rescue drugs used | Within postoperative 24 hours
The incidence of postoperative hypotension and bradycardia | From the administration of experimental drugs to postoperative 24 hours
Ramsay sedation score | Within postoperative 3 days
  The minimum and maximum score are 1 and 6, respectively. Score 1 represents that patients is anxious and agitated or restless , or both. And score 6 represents that patients exhibits no response.
Postoperative extubation time | The time of extubation
Length of stay in the ICU | The length of stay in ICU within postoperative 30 days
The incidence of postoperative delirium | Within postoperative 7 days
The incidence of postoperative arrhythmias | Within postoperative 24 hours
The incidence and severity of postoperative PONV | Within postoperative 3 days
Length of stay | The first day after surgery to discharge
The rate of all-cause death of participants | Within postoperative 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- China, Shandong Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao C, Lv M, Wei C, Yan J, Wang Y, Gu C. Comparison of dexmedetomidine and meperidine for the prevention of shivering following coronary artery bypass graft: study protocol of a randomised controlled trial. BMJ Open. 2022 Feb 11;12(2):e053865. doi: 10.1136/bmjopen-2021-053865. PMID 35149565